CLINICAL TRIAL: NCT06933498
Title: Comparison of the Effects of Preoperative and Intraoperative Erector Spinae Plane Block on Opioid Consumption, Anesthetic Consumption and Hemodynamics in Lumbar Disc Herniation Surgeries.
Brief Title: Effects of Erector Spinae Plane Block on Opioid Consumption, Anesthetic Consumption and Hemodynamics in Lumbar Disc Herniation Surgeries.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, Clinic Associate Professor, Ankara Ataturk Sanatorium Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-KAEK-24/14
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Erector Spina Plan Block; Opioid Consumption; Postoperative Pain
Keywords: Lumbar disc herniation surgery.; Erector spinae plane block; Anesthetic drug consumption; Opioid consumption; Perioperative hemodynamics
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients who volunteer to participate in the study will be randomly assigned to the patient groups that will receive preoperative ESPB and intraoperative ESPB in a 1:1 ratio. This process will be performed using a computer-based program that follows a random number generator protocol. Patients will be classified using the online calculator at www.calculator.net. A random number will be assigned to each patient according to the calculator output. The group to be applied preoperative ESPB will include patients between numbers 1 and 30, and the group to be applied intraoperative ESPB will include patients between numbers 31 and 60.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PREOPERATİVE ESPB (Active Comparator): After 0.03 mg/kg IV midazolam sedation is applied to patients who will undergo preoperative ESPB, bilateral ultrasound-guided ESPB (in-plane approach) will be applied over the vertebral level that is equidistant from the highest and lowest vertebral levels planned for surgery in the prone position. ESPB will be performed by experienced anesthesiologists. After sterilization of the skin with povidone iodine, the probe with a sterile sheath is placed 3 cm lateral to the spinous process and the trapezius, rhomboid major, erector spinae muscles and the transverse process of the vertebrae are visualized. The needle is placed in the fascial plane on the deep surface of the erector spinae muscle on the bone shadow of the transverse process of the vertebra. A total of 40 mL of 0.25% bupivacaine is administered bilaterally after the LA spread is seen. After waiting for the effect of the block for 30 minutes, the patients will be taken to the operating room.
  Interventions: Procedure: PREOPERATIVE ESPB
- INTRAOPERATİVE ESPB (Active Comparator): Intraoperative ESPB will be performed by the neurosurgeon after LDH repair, starting from the level of the operated vertebra and covering all surgical segments. This procedure will be repeated for the other side (right/left). A total of 40 mL of 0.25% bupivacaine will be used for both sides.
  Interventions: Procedure: INTRAOPERATIVE ESPB

INTERVENTIONS:
Procedure: PREOPERATIVE ESPB — After 0.03 mg/kg IV midazolam sedation is applied to patients who will undergo preoperative ESPB, bilateral ultrasound-guided ESPB (in-plane approach) will be applied over the vertebral level that is equidistant from the highest and lowest vertebral levels planned for surgery in the prone position. ESPB will be performed by experienced anesthesiologists. After sterilization of the skin with povidone iodine, the probe with a sterile sheath is placed 3 cm lateral to the spinous process and the trapezius, rhomboid major, erector spinae muscles and the transverse process of the vertebrae are visualized. The needle is placed in the fascial plane on the deep surface of the erector spinae muscle on the bone shadow of the transverse process of the vertebra. A total of 40 mL of 0.25% bupivacaine is administered bilaterally after the LA spread is seen. After waiting for the effect of the block for 30 minutes, the patients will be taken to the operating room.
  Arms: PREOPERATİVE ESPB
Procedure: INTRAOPERATIVE ESPB — Intraoperative ESPB will be performed by the neurosurgeon after LDH repair, starting from the level of the operated vertebra and covering all surgical segments. This procedure will be repeated for the other side (right/left). A total of 40 mL of 0.25% bupivacaine will be used for both sides.
  Arms: INTRAOPERATİVE ESPB

SUMMARY:
Lumbar disc herniation (LDH) is an increasingly common spine disorder . In patients treated surgically, inhalation anesthesia and the use of opioids for analgesic purposes are generally the chosen anesthetic methods. Surgical techniques such as discectomy, microdiscectomy, and stabilization (REF) are used to treat LDH. Although discectomy is considered the primary option in the treatment of LDH, less invasive techniques such as microdiscectomy have been applied in recent years . However, despite the use of less invasive techniques, patients experience pain after surgery . Clinicians want to avoid complications such as thromboembolism and hemodynamic deterioration that may occur due to postoperative pain, and to apply effective pain treatment for patient comfort and rapid discharge from the hospital. It has also been stated that inadequate postoperative pain treatment may increase the risk of developing chronic pain. Therefore, the use of opioids for analgesic purposes in the intraoperative and postoperative periods is quite common. However, opioid use may cause side effects that negatively affect postoperative recovery and may delay discharge. Some of these situations include delayed recovery from anesthesia, failure to perform early postoperative neurological examination due to delayed recovery, postoperative nausea and vomiting (PONV), pruritus, urinary retention, respiratory depression, gastrointestinal dysfunction, and addiction.

Another important issue is the difficulty of applying effective treatment to patients, the side effects that develop due to the applied treatments, and the increase in healthcare costs, which are important problems. Therefore, it is also very important to take a cost-effective approach while trying to treat patients at the highest level. The applied anesthesia and analgesia methods can also significantly affect the cost of surgical treatments. In particular, inhalation anesthetics used in patients receiving general anesthesia and opioids used for intraoperative and postoperative analgesia constitute a significant portion of the anesthesia cost. Therefore, strategies that will provide cost savings by reducing the use of both inhalation anesthetics and opioids are emphasized. In this context, nerve blocks or fascial plane blocks applied with local anesthetics come to the fore. With the widespread use of ultrasonography in regional anesthesia practice, regional plane blocks have also become widespread in parallel with this development and have begun to take more place in the literature. Erector spinae plane block (ESPB) is also among these blocks that are increasingly gaining ground in the literature. ESPB is a technique defined for both acute and chronic pain. ESPB is performed by administering local anesthetic (LA) to the fascial plane between the transverse process of the vertebra and the overlying erector spinae muscle. When literature data are examined, ESPB can be applied from the thoracic or lumbar levels in LDH surgery, before and after preoperative anesthesia induction, intraoperatively, at the end of surgery, before extubation or in the postoperative period. ESPB can be applied with the patient in the prone position, sitting or lateral decubitus position.

In studies conducted on patients undergoing laparoscopic cholecystectomy, it was found that ESPB reduced the amount of intraoperative inhalation anesthetic and opioid consumption. In another study examining the effect of ESPB on lumbar spine surgeries, it was found that ESPB reduced the use of intraoperative fentanyl and isoflurane and significantly shortened the recovery time. In addition, ESPB is thought to provide more effective analgesia in postoperative pain management and reduce opioid consumption and opioid-related side effects after lumbar spine surgeries. According to the results of published studies, it has been stated that ESPB is more effective for postoperative analgesia in patients undergoing lumbar surgery, significantly reduces pain scores at rest (static) and during activity (dynamic), provides a significant decrease in 24-hour opioid consumption, prolongs the first analgesic requirement period and is associated with fewer side effects.

Another important issue is to keep intraoperative hemodynamics stable within normal limits in patients under general anesthesia. Hemodynamic stability is very important to ensure that the amount of bleeding from the surgical site is kept at a minimum level, especially during LDH surgeries. It has been stated that the combined application of regional anesthesia and general anesthesia in spinal surgery provides better pain control as well as better hemodynamic stability.

This study aimed to compare the effects of preoperative and intraoperative ESPB on opioid consumption, anesthetic drug consumption, and hemodynamics in LDH surgeries.

DETAILED DESCRIPTION:
This thesis study will be conducted in accordance with the Declaration of Helsinki and will be conducted at SBÜ Ankara Atatürk Sanatoryum Education and Research Hospital

Patients between the ages of 18-75 who will undergo surgery due to LDH and who agree to participate in this study and sign the informed consent form will be prospectively recorded. A total of 60 patients will be included in our study. All patients will be informed about the process and their informed consent will be obtained.

The standard anesthesia and analgesia protocol that we routinely apply will be applied to the patients throughout the surgery. Patients who volunteer to participate in the study will be randomly assigned to the patient groups that will receive preoperative ESPB and intraoperative ESPB in a 1:1 ratio. This process will be performed using a computer-based program that follows a random number generator protocol. Patients will be classified using the online calculator at www.calculator.net. A random number will be assigned to each patient according to the calculator output. The group to be applied preoperative ESPB will include patients between numbers 1 and 30, and the group to be applied intraoperative ESPB will include patients between numbers 31 and 60.

The list created will be kept in a locked file to be used by the clinical research team at the beginning of the study. This method will ensure that randomization is unbiased and equally distributed between the groups.

All patients will be given standard multimodal analgesia in the postoperative period. At the end of the study, the data of the patient groups to which preoperative ESPB and intraoperative ESPB were applied will be compared according to the time of ESPB.

If the patient has pain after the surgery, the patient will not wait and the necessary analgesic treatment will be given to the patient. Demographic data of the patients (age, height, body weight, BMI, gender), preoperative routine blood tests, diagnoses, ASA score, preoperative VAS score, type of surgery performed, duration of surgery, complications if any developed during the procedure or postoperative follow-up, hemodynamic data before anesthesia induction, after induction, at the 5th, 10th, 15th, 20th, 25th, 30th, 35th, 40th, 45th, 60th, 90th, 105th and 120th minutes of intubation, just before extubation, after extubation (systolic arterial pressure (SAB), diastolic arterial pressure (DAB), mean arterial pressure (MAP), heart rate (HR), peripheral oxygen saturation (SpO2) will be recorded. Sevoflurane minimum alveolar concentration (MAC) values will also be recorded at the same measurement times. Total amount of inhaled anesthetic used during the intraoperative period, intraoperative opioid consumption, postoperative 1st, 2nd, 4th, 8th, 16th, 24th, 36th and 48th hours at rest and during movement will be recorded on the Visual Analog Scale (VAS). Total postoperative opioid consumption and additional analgesic requirement will also be recorded. During the VAS evaluation, the patient will be asked to show the location of the pain when evaluated on a 100 mm scale as 0: no pain, 100: maximum pain, and the value shown by the patient will be recorded.

During this process, side effects such as dizziness, nausea-vomiting, hypotension, bradycardia, itching, sweating, and respiratory depression due to pain treatment will be recorded.

GENERAL ANESTHESIA MANAGEMENT All patients will be monitored according to ASA monitoring standards. According to our general anesthesia protocol, after premedication with 0.03 mg/kg intravenous (i.v.) midazolam, propofol 2-2.5 mg/kg (i.v.) and fentanyl 1-1.5 mg/kg (i.v.) and 0.6 mg/kg (i.v.) rocuronium will be administered for anesthesia induction. Anesthesia will be maintained with controlled ventilation at 2 L fresh gas (FG) flow with 2% sevoflurane in a mixture of 50% air and 50% oxygen. The depth of anesthesia will be monitored by keeping the bispectral index (BIS) (COVIDIEN) score between 40-60, and increasing or decreasing sevoflurane concentration will be provided according to the depth of anesthesia. Remifentanil (0.5-1 μg/kg/min) infusion will be applied to ensure adequate depth of anesthesia and hemodynamic stability. For postoperative analgesia, our standard analgesia protocol will be applied to patients 30 minutes before the end of the surgical procedure. After adequate muscle strength and spontaneous ventilation are achieved with 2-4 mg/kg sugammadex, patients will be extubated and transferred to the postoperative recovery unit.

Sevoflurane application time and concentration, constant fresh gas (FG) flow will be recorded. The total amount of sevoflurane consumption at the end of the surgery will be determined from these records.

ERECTOR SPINA PLAN BLOCK After 0.03 mg/kg IV midazolam sedation is applied to patients who will undergo preoperative ESPB, bilateral ultrasound-guided ESPB (in-plane approach) will be applied over the vertebral level that is equidistant from the highest and lowest vertebral levels planned for surgery in the prone position. ESPB will be performed by experienced anesthesiologists. After sterilization of the skin with povidone iodine, the probe with a sterile sheath is placed 3 cm lateral to the spinous process and the trapezius, rhomboid major, erector spinae muscles and the transverse process of the vertebrae are visualized. The needle is placed in the fascial plane on the deep surface of the erector spinae muscle on the bone shadow of the transverse process of the vertebra. A total of 40 mL of 0.25% bupivacaine is administered bilaterally after the LA spread is seen. After waiting for the effect of the block for 30 minutes, the patients will be taken to the operating room.

Intraoperative ESPB will be performed by the neurosurgeon after LDH repair, starting from the level of the operated vertebra and covering all surgical segments. This procedure will be repeated for the other side (right/left). A total of 40 mL of 0.25% bupivacaine will be used for both sides.

Standard analgesia protocol will be applied for postoperative analgesia in both groups where ESPB is applied.

STANDARD POSTOPERATIVE ANALGESIA PROTOCOL 30 minutes before the end of the surgical procedure, patients will be given IV dexketoprofen (50 mg), tramadol (100 mg), and metoclopramide to prevent nausea and vomiting. In the postoperative period, intravenous morphine will be administered via a patient-controlled analgesia (PCA) pump for 24 hours. Pain intensity will be assessed using a 100-point (0: No pain and 100: Unbearable pain) VAS. The dose delivery of the PCA pump will be limited to administering a 1 mg morphine bolus dose and delivering a maximum total dose of 12 mg morphine over 4 hours with 15-minute lockout intervals. For multimodal analgesia, 1 g paracetamol every 8 hours and 50 mg dexketoprofen twice daily will be administered intravenously. As a rescue analgesic agent, 0.5 mg/kg tramadol will be administered intravenously to patients when the VAS score is ≥ 40. VAS scores will be recorded at postoperative 1st hour, 2nd hour, 4th hour, 8th hour, 16th hour, 24th hour, 36th hour and 48th hour.

ELIGIBILITY:
Inclusion Criteria:

* Those over 18 and under 75 years of age,
* Those with an American Society of Anesthesiologists (ASA) score of I-II-III,
* Those with a body mass index (BMI) between 18-40 kg/m2
* Patients undergoing surgery with general anesthesia
* Patients undergoing LDH surgery (levels 1, 2, and 3)
* Patients with informed consent

Exclusion Criteria:

* Patients with severe cardiovascular system disease,
* Patients with coagulation disorders,
* Those allergic to the anesthetic and analgesic drugs to be administered,
* Patients with infection at the injection site,
* Patients with severe renal failure, gastrointestinal ulceration or severe asthma that prevents standard analgesia protocol
* Patients who have previously undergone LDH surgery at the same level,
* Patients who are planned to have surgery at more than 3 levels
* Patients with ASA 4 and above,
* Patients who are planned with total intravenous anasthesia(TIVA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 24 hours
  The total amount of morphine consumption
anesthetic consumption | 24 hours
  The total amount of sevoflurane consumption at the end of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Karabulut, Principal Investigator — Ankara Atatürk Sanatorium Training and Research Hospital Recruiting Ankara, Keçiören, Turkey
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No